CLINICAL TRIAL: NCT00268125
Title: Evaluation of Acupression's Bracelets Associated to an Educational Step Versus Education Only in Nausea and Vomiting's Mastering Induced by FEC100 Chemotherapy's Sort.
Brief Title: Phase 3 Study of Acupression's Bracelets in Nausea and Vomiting Induced by FEC100 Chemotherapy's Sort.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Dr Jean-Pierre DELORD, Institut Claudius Regaud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05 DIVE 05
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasm; FEC100; Chemotherapy; acupression; bracelet; nausea; vomiting
MeSH Terms: conditions — Breast Neoplasms; Nausea; Vomiting | interventions — Hygiene

INTERVENTIONS:
Device: Acupression's bracelet
Behavioral: Hygiene and dietetic advices

SUMMARY:
The purpose of this study is to demonstrate a betterment of the digestive symptomatology by the anti-emetic acupression's bracelets's use associated with hygiene and dietetic advices.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Age > 18 years
* Well-informed written consent, signed by the patient before the beginning of the study
* Breast cancer's diagnosis (operated or not)
* Forecast of a treatment by FEC100 chemotherapy's sort (D1=D21) during at least 3 cycles.
* Patient affiliated at a welfare or beneficiary from it
* Investigator estimates that the patient is able to conform with protocol's conditions and to respect them

Exclusion Criteria:

* Operated arm's lymphedema
* Wrist's morphology which cannot permit the bracelet's wearing (20 cm)
* D1=D15 FEC100's treatment
* Psychic incapability to sign a well-informed consent
* Refusal to give a written consent
* Patient under tutelage or guardianship
* Pregnant or breast-feeding woman
* Any clinical trial's participation which would impose nausea and vomiting's treatment modalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 347 (Estimated)
Dates: Start 2006-02; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Reduction of 15% of stage III/IV nausea and vomiting's incidence.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre DELORD, Dr, Principal Investigator — Institut Claudius Regaud
Locations (3):
- France (3):
  - Centre Oscar Lambret, Lille
  - Centre Paul STRAUSS, Strasbourg
  - Institut Claudius Regaud, Toulouse